CLINICAL TRIAL: NCT00038896
Title: A Double-blind, Placebo-controlled, Parallel-group, Flexible-dose Study of Venlafaxine Extended-release Capsules in Adult Outpatients With Panic Disorder
Brief Title: Study Evaluating Venlafaxine ER in Adults With Panic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0600B5-353
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Panic Disorder
Keywords: Panic; Disorder
MeSH Terms: conditions — Panic Disorder; Disease

INTERVENTIONS:
Drug: Venlafaxine ER

SUMMARY:
The primary objective of this study is to determine the efficacy, safety, and tolerability of a flexible dose of venlafaxine extended-release (ER) capsules administered for 10 weeks in the treatment of adult outpatients with panic disorder (PD) in a placebo-controlled phase III study.

ELIGIBILITY:
Inclusion Criteria:

* A male or female outpatient
* Be at least 18 years of age and legal age of consent
* Meet DSM-IV criteria for PD (with or without agoraphobia) for at least 3 months before study day 1

Exclusion Criteria:

* Treatment with venlafaxine (IR or ER) within 6 months of study day 1
* Known hypersensitivity to venlafaxine (IR or ER) or related compounds
* History or presence of any clinically important hepatic, renal, or other medical disease that might compromise the study or be detrimental to the patient (eg, clinically important cardiac arrhythmia, unstable diabetes, carcinoma [except basal cell epithelioma], uncontrolled hypertension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2001-04; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Liebowitz MR, Asnis G, Mangano R, Tzanis E. A double-blind, placebo-controlled, parallel-group, flexible-dose study of venlafaxine extended release capsules in adult outpatients with panic disorder. J Clin Psychiatry. 2009 Apr;70(4):550-61. doi: 10.4088/jcp.08m04238. Epub 2009 Apr 7. PMID 19358784